CLINICAL TRIAL: NCT02754934
Title: Development of a Self-administered Neck Mobility Assessment Tool in Chronic Neck Pain Patients.
Status: Completed | Type: Observational
Sponsor: Balgrist University Hospital (Other)
Collaborators: Maastricht University (Other)
Responsible Party: Principal Investigator, Swanenburg, Senior Researcher, Balgrist University Hospital
Other Study IDs: 2016-00164
Record Dates: First submitted 2016-04-25; First posted 2016-04-28 (Estimated); Last update posted 2016-11-04 (Estimated); Status verified 2016-11

CONDITIONS: Neck Pain
Keywords: chronic
MeSH Terms: conditions — Neck Pain; Bronchiolitis Obliterans Syndrome

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Cervical range of motion — Patients will fill out the Neck Disability Index, Visual Analogue Pain Rating Scale and the Self-administered Neck range of motion questionnaire.

SUMMARY:
This study evaluates, if the movement of the cervical spine, assessed via a specific questionnaire by the patient, is a valid and reliable tool and could be used in daily clinical routine.

DETAILED DESCRIPTION:
Cervical range of motion is a frequently used assessment methods in patients with neck pain.

Although it seems to be used frequently, clinicians still prefer hands-on assessment. Furthermore it is interesting, if cervical range of motion,self-assessed by the patient is a valid and reliable tool.

ELIGIBILITY:
Inclusion Criteria:

* Neck pain > 90 days
* Able to speak, read and write German

Exclusion Criteria:

* Red Flags e.g. Fracture of the cervical spine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Investigators will include 50 participants with chronic neck pain
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2014-11; Primary Completion 2016-09 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Cervical Spine Mobility | Day one of the study
  Patients will fill out the questionnaire once, at the beginning of the study.

SECONDARY OUTCOMES:
Pain Visual Analogue Pain Rating Scale | Day one of the study
  Patients will fill out the questionnaire once, at the beginning of the study.
Disability on Neck Disability Index | Day one of the study
  Patients will fill out the questionnaire once, at the beginning of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Jaap Swanenburg, PhD, Principal Investigator — Balgrist University Hospital
Locations (1):
- Balgrist University Hospital, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Langenfeld A, Bastiaenen C, Sieben J, Swanenburg J. Development and validation of a self-administered neck mobility assessment tool (S-ROM-Neck) in chronic neck pain patients. Musculoskelet Sci Pract. 2018 Oct;37:75-79. doi: 10.1016/j.msksp.2018.04.004. Epub 2018 Apr 10. PMID 29656846